CLINICAL TRIAL: NCT06798623
Title: Anterior Cruciate Ligament (ACL) Reconstruction With Autologous Fat Pad Derived Mesenchymal Stem Cells
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Patrick McCulloch,MD, John S. Dunn Chair in Orthopedic Surgery, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00039160
Record Dates: First submitted 2025-01-20; First posted 2025-01-29 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intra-articular injection of autologous mesenchymal stromal cells (Experimental): Each subject will receive one intra-articular injection of autologous mesenchymal stromal cells derived from infrapatellar fat pad (FP-MSC) tissue samples collected from the subject during anterior cruciate ligament (ACL) reconstruction surgery.
  Interventions: Biological: Autologous Mesenchymal Stromal Cells

INTERVENTIONS:
Biological: Autologous Mesenchymal Stromal Cells — Autologous mesenchymal stromal/stem cells extracted from the subject during a routine standard of care ACL reconstruction surgery and reintroduced in one clinic visit approximately 21 days after completion of the surgery. After being removed from the patient, the cells will be cultured, modified, and harvested to become the final investigational product. Each subject will receive 1.5 ml of the investigative drug. This will contain 5x10^7 (50 million) autologous MSCs.

SUMMARY:
This study is designed as a prospective, open label, single arm pilot clinical study that will establish the safety and efficacy of a single injection of mesenchymal stromal cells in patients. Each subject will receive one intra-articular injection of autologous mesenchymal stromal cells derived from infrapatellar fat pad (FP-MSC) tissue samples collected from the subject during anterior cruciate ligament (ACL) reconstruction surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older who are scheduled to undergo anterior cruciate ligament (ACL) reconstruction with the Principal Investigator (PI).
* Receiving post-surgery physical therapy at a Houston Methodist physical therapy (PT) clinic.

Exclusion Criteria:

* Under 18 years of age
* Prior surgery on affected knee
* Diabetes
* Root repair, inflammatory arthropathy, or any other concomitant procedure that cannot follow an accelerated PT protocol or any concomitant procedure that the PI deems exclusionary
* Unable to attend physical therapy at Houston Methodist
* Vulnerable populations
* Immunocompromised patients such as those being treated for cancer, kidney failure, etc.
* Heart disease including (systolic blood pressure >180 mm Hg or heart failure)
* Active infections
* Non-English-speaking patients
* Any known metal implants or allergy to contrast agents
* Pregnancy (as part of standard of care, all female participants will be administered a urine pregnancy test prior to surgery. A negative result is required to proceed with surgery per SOC and thus, participate in the study) and those planning to become pregnant during the duration of the study
* Any condition with known bleeding disorders, thrombus formation risk factors, or overlying wound and skin infections
* Any condition in the opinion of the primary investigator that would compromise the integrity of the data collection or outcomes being assessed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 4-5 weeks postop, 6-7 weeks postop, 3.5 months postop, 6 months postop
  Participants will be asked via a follow-up phone call following injection whether or not they have experienced any adverse events following the injection. They will be assessed at all remaining standard of care follow up visits and staff will inquire about adverse events.
Knee Function | Preoperative appointment, 6 weeks postop, 3.5 months postop, 6 months postop
  Knee function will be assessed through patient reported responses on the Knee Injury and Osteoarthritis Outcome Score (KOOS) survey via REDCap. The Questionnaire has five subscales which are separately scored (pain, function in daily living, function in sport and recreation, other symptoms and knee-related quality of life). Final score will be determined on a scale of 0-100 where 100 indicates no symptoms and 0 indicates extreme symptoms.
Knee Function | Preoperative appointment, 6 weeks postop, 3.5 months postop, 6 months postop
  Function will be assessed with the International Knee Documentation Committee Subjective Knee Form (IKDC) which contains sections on knee symptoms, function, and sports activities. Total score will range from 0 (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Knee Function | Preoperative appointment, 6 weeks postop, 3.5 months postop, 6 months postop
  Active and passive Range of Motion (ROM) of the operated and contralateral knee will be documented by the physician. This will be determined by the measurement of angles in each plane at the body's joints.

SECONDARY OUTCOMES:
Knee Pain | Preoperative appointment, 6 weeks postop, 3.5 months postop, 6 months postop
  Pain levels will be assessed using patient reported outcomes via REDCap. The Visual Analogue Scale will ask participants to mark on a line, using a ruler, how much pain they are in. The score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Return to Sport Time | 3 months postop
  Return to sport time will be evaluated via the subject's standard of care (SOC) physical therapy notes in their chart.
Knee Swelling | Preoperative appointment, 6 weeks postop, 3.5 months postop, 6 months postop
  The trans-patellar circumference of both knees will be measured at the standard of care (SOC) appointments the subject will attend throughout the study to monitor swelling. Knees will be measured utilizing a flexible measuring tape and the affected knee will be compared to the unaffected knee to verify the difference in size, and therefore the severity of swelling. The greater the difference in size between knees, the more severe the swelling.
Knee Pain | Preoperative appointment, 6 weeks postop, 3.5 months postop, 6 months postop
  Questions related to pain will also be assessed on the International Knee Documentation Committee Subjective Knee Form (IKDC), although this is not its primary focus. Total score will range from 0 (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick McCulloch, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No